CLINICAL TRIAL: NCT05135715
Title: A Single-arm, Multicentre, Open Phase Ⅱa Clinical Study of RC48-ADC in the Treatment of HER2 Variant (Mutation, Amplification, Overexpression) Advanced Melanoma
Brief Title: A Study of RC48-ADC in Advanced Melanoma Subjects With HER2 Variant (Mutation, Amplification, Overexpression)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C020
Record Dates: First submitted 2021-11-15; First posted 2021-11-26 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-11

CONDITIONS: Melanoma, Stage II; HER2-positive; Advanced Melanoma
Keywords: RC48-ADC; HER2-positive melanoma
MeSH Terms: conditions — Melanoma | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48-ADC (Experimental): Participants will receive RC48-ADC every 2 weeks (Q2W) until investigator assessed loss of clinical benefit, unacceptable toxicity, investigator or participant decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: RC48-ADC

INTERVENTIONS:
Drug: RC48-ADC — 2.0 mg/kg IV every 2 weeks
  Other Names: Recombinant Humanized anti-HER2 Monoclonal Antibody-MMAE Conjugate For Injection

SUMMARY:
This is a Phase IIa, single-arm, multicentre, open-label clinical trial aims to evaluate the effectiveness and safety of RC48-ADC in the treatment of HER2 Variant (Mutation, Amplification, Overexpression) advanced melanoma.

DETAILED DESCRIPTION:
This study is a phase IIa multicentre,single-arm, open-label, clinical study to evaluate the efficacy and safety of recombinant humanized anti-HER2 monoclonal antibody-Monomethyl auristatin E (MMAE) conjugate for the treatment of HER2- positive advanced melanoma. HER2 mutation is defined as the presence of HER2 gene mutations in primary or metastatic tumour tissue as detected by immunohistochemistry (IHC). HER2 gene mutation.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent.
* Male or female, Age ≥ 18 years.
* Predicted survival ≥ 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* All female subjects will be considered to be of child-bearing potential unless participants are postmenopausal, or have been sterilized surgically.Female subjects of child-bearing potential must agree to use two forms of highly effective contraception. Male subjects and their female partner who are of child-bearing potential must agree to use two forms of highly effective contraception.
* Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.
* Adequate organ function.
* All subjects must be histologically confirmed, non-resectable stage III or metastatic melanoma, except for patients with uveal or ocular melanoma.
* The subject has experienced disease progression or intolerance after receiving standard treatment in the past; Patients with disease progression within 6 months after receiving neoadjuvant or adjuvant chemotherapy regimens can be included in the clinical study.
* The HER2 IHC test result is IHC 2+ or IHC 3+, the subject's previous test results (confirmed by the investigator) or the research center's test results are acceptable; the subject can provide the Specimen of primary or metastatic tumor for HER2 review/judgment.
* According to the RECIST 1.1 standard, there is at least one measurable lesion.

Exclusion Criteria:

* Known hypersensitivity to Recombinant Humanized Anti-HER2 Monoclonal Antibody-MMAE Conjugate For Injection.
* History of receiving any anti-cancer drug/biologic treatment within 4 weeks prior to trial treatment.
* Pleural or abdominal effusion with clinical symptoms that requires ongoing treatment.
* Treated with systemic treatment (e.g. immunomodulators, corticosteroids or immunosuppressants) for the autoimmune disease within 2 years prior to the study treatment.
* History of major surgery within 4 weeks of planned start of trial treatment.
* Has received a live virus vaccine within 4 weeks of planned start of trial treatment.
* Toxicity of previous anti-tumor treatment not recovered to CTCAE Grade 0-1 (with exception of Grade 2 alopecia).
* Pregnancy or lactation.
* Currently known active infection with HIV or tuberculosis.
* Diagnosed with HBsAg, HBcAb positive and HBV DNA copy positive, or HCVAb positive.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or cancers with a similar curative outcome as those mentioned above.
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate (ORR) | within approximately 3 years
  The objective response rate will be analyzed according to the RECIST 1.1 standard tumor evaluation.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | within approximately 3 years
  Progression-free survival (PFS) refers to the time from the date of randomization to the first researcher's evaluation of disease progression or death (calculated by the event that occurred first). The disease progression will be evaluated by the researchers according to the RECIST 1.1 standard.
Duration of relief (DOR) | within approximately 3 years
  DOR is defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death.
Disease control rate (DCR) | within approximately 3 years
  Disease control rate (DCR) is defined as cases where objective remission (assessed as complete remission or partial remission according to RECIST 1.1 standard) or stable disease during the study.
Overall survival (OS) | within approximately 3 years
  Overall survival (OS) refers to the time from the date of randomization to the date of death of the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, Ph.D, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (4):
- China (4):
  - Fujian cancer hospital, Fuzhou, Fujian
  - The First Hospital of Jilin University, Changchun, Jilin
  - Zhejiang cancer hospital, Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing